CLINICAL TRIAL: NCT04662723
Title: Multicentre Prospective Open Label Clinical Study to Evaluate the Effect of Personalized Therapy on Patients With Immunoglobulin A Nephropathy.
Brief Title: Multicentre Clinical Study to Evaluate the Effect of Personalized Therapy on Patients With Immunoglobulin A Nephropathy.
Acronym: CLIgAN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Schena (Other)
Collaborators: University of Bari (Other)
Responsible Party: Principal Investigator, Francesco Paolo Schena, President and scientif director, Fondazione Schena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2020-11-27; First posted 2020-12-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Glomerulonephritis; Immunoglobulin A Nephropathy
Keywords: IgA nephropathy; Steroids; RAS-blockers; SGLT2-inhibitors
MeSH Terms: conditions — Glomerulonephritis; Glomerulonephritis, IGA | interventions — Adrenal Cortex Hormones; Methylprednisolone Hemisuccinate; Prednisolone; Ramipril; Lisinopril; Losartan; Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin; Canagliflozin; empagliflozin

STUDY DESIGN:
Intervention Model Description: After the enrolment the eligible biopsy-proven IgAN patients will be randomized, separately, in each trial in a 1 to 1 ratio via a web-based program generating random numbers. The allocation will be not blinded to the group of assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Corticosteroids combined with RASBs (Experimental): Patients assigned to the corticosteroid group will receive (pulse) methylprednisolone succinate 500-1000 mg/day for 3 consecutive days followed by oral prednisolone (0.5 mg/kg/bw) on alternate days until the end of month. This treatment will be repeated for three consecutive months. In addition, patients will receive RASBs that will be titrated to their maximum anti-proteinuric effect. The dose of methylprednisolone succinate will be individualized (15 mg/kg) based on the ideal body weight. In overweight and obese IgAN patients the ideal body weight will be considered. The drug will be administered in a single daily dose intravenously for 30-60 min. To avoid obesity and diabetes corticosteroids will be administered only in the morning.
  Interventions: Drug: Corticosteroid; Drug: Renin-angiotensin sytem blockers
- RASBs (Active Comparator): Patients will receive RASBs for 3 months, titrated to their maximum anti-proteinuric effectf followed by oral corticosteroids.
  Interventions: Drug: Renin-angiotensin sytem blockers
- SGLT2i combined with Ramipril (Experimental): IgAN patients with chronic renal lesions (T1,2) or moderate renal lesions (M0,1; S0,1; T0; E0; C0) at high or very high CKD risk (proteinuria> 0.5 g/day and GFR >30ml/min/1.73 m2) will receive SGLT2i combined with RASBs.
  Interventions: Drug: Renin-angiotensin sytem blockers; Drug: Sodium-glucose cotransporter 2 inhibitor
- Ramipril combined with corticosteroids (Active Comparator): IgAN patients with chronic renal lesions (T1,2) or moderate renal lesions (M0,1; S0,1; T0; E0; C0) at high or very high CKD risk (proteinuria> 0.5 g/day and GFR >30ml/min/1.73 m2) will receive RASBs for 3 months followed by oral corticosteroids.
  Interventions: Drug: Corticosteroid; Drug: Renin-angiotensin sytem blockers

INTERVENTIONS:
Drug: Corticosteroid — To reduce the progression of renal damage in IgAN Patients
  Other Names: Methylprednisolone succinate; prednisolone
  Arms: Corticosteroids combined with RASBs; Ramipril combined with corticosteroids
Drug: Renin-angiotensin sytem blockers — To reduce the progression of renal damage in IgAN Patients
  Other Names: Ramipril; lisinopril; losartan
Drug: Sodium-glucose cotransporter 2 inhibitor — To reduce the progression of renal damage in IgAN Patients
  Other Names: dapagliflozin; canagliflozin; empagliflozin
  Arms: SGLT2i combined with Ramipril

SUMMARY:
Idiopathic immunoglobulin A nephropathy (IgAN) is the most common biopsy-proven glomerulonephritis in the world. Approximately 40% of IgAN patients reach end-stage kidney disease (ESKD) 20 years after their kidney biopsy. The high prevalence of ESKD suggests the need to move from a generalized therapy for all patients to personalized therapy.

Many RCTs have been conducted stratifying patients based on the laboratory findings (serum creatinine, eGFR and daily proteinuria). In contrast, data from the kidney biopsy has been used only for clinical diagnosis. Therefore, IgAN patients with active or chronic renal lesions have not been equally distributed in experimental and control arms of the randomized clinical trials (RCTs) Our clinical study of IgAN (CLIgAN) is a multicentre, prospective, controlled and open-label randomized clinical trial based on patients' stratification at the time of their kidney biopsy. The investigators will consider, first, the type of renal lesions followed by the serum creatinine values, eGFR and proteinuria. IgAN patients with active renal lesions (n=132) will be enrolled in the first RCT (ACIgAN) in which they will receive corticosteroids (pulse therapy) plus oral corticosteroids combined with RASB or RASB followed by oral corticosteroids. IgAN patients with chronic or moderate renal lesions at high or very high risk of chronic renal disease (n=294) will be enrolled in the second RCT (CHRONIgAN) in which they will receive the SGLT2 inhibitor combined with RASB compared with RASB combined with oral corticosteroids. Using this approach, the investigators hypothesize that patients could receive personalized therapy based on renal lesions to ensure that the right drug gets to the right patient at the right time.

Recently, we developed a Clinical Decision Support System (CDSS) tool using artificial intelligence (artificial neural networks) to identify IgAN patients at high risk of developing ESKD. The IgAN tool (DialCheck) was validated in a retrospective cohort of IgAN patients but not in a prospective clinical study. The investigators propose to measure the power of the DiaCheck tool in patients enrolled in both RCTs to determine whether personalized therapy can slow the decline of the renal function to delay the ESKD.

The CLIgAN study also includes a cutting-edge molecular study for precision therapy (PRECIgAN).

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE. Idiopathic Immunoglobulin A nephropathy (IgAN) is the most common biopsy-proven glomerulonephritis in the world. It is more prevalent in Asia than in Europe and the US. Approximately 40% of IgAN patients reach end-stage kidney disease (ESKD) 20 years after their kidney biopsy. The high prevalence of ESKD shows that IgAN has a significant economic impact in the all countries because renal replacement therapy is costly. Moreover, the disease's onset in the second and third decades of life represents a social challenge because young adult patients are very active and highly productive in the workplace. This challenge is one more reason to move from a generalized therapy for all patients to a personalized therapy.

The first edition of the KDIGO guidelines, published in 2012, suggested different therapeutic approaches for IgAN patients based on the clinical setting. However, the KDIGO guidelines do not consider the presence of active (endocapillary and extracapillary lesions) and chronic (tubulointerstitial lesions) renal lesions at the time of the kidney biopsy for therapy decision. The investigators of the clinical study in IgAN patients (CLIgAN) will consider for the patient's stratification the type of renal lesions, preliminarily, and then the clinical parameters as estimated glomerular filtration rate (eGFR) and proteinuria because the categorization of proteinuria and eGFR is not enough for a complete diagnosis of the disease.

AIMS. Considering the critical role of kidney biopsy, in the CLIgAN study the investigators plan to evaluate (i) the effect of corticosteroids combined with RASBs in IgAN patients with active renal lesions (ACIgAN) versus RASBs for 3 months followed by oral corticosteroids to determine whether the renal lesions are reversed by immediate corticosteroid therapy; (ii) the effect of SGLT2i in patients with chronic or moderate renal lesions (CHRONIgAN) to determine whether a delay of the ESKD onset is achieved; (iii) after the prediction of ESKD through the IgAN CDSS tool (DialCheck), to determine whether personalized therapy delays the impairment of the renal function; (iv) finally, on a small cohort of active and chronic IgAN patients enrolled in the CLIgAN study, a cutting edge-molecular study will be conducted to evaluate the effect of precision therapy (PRECIgAN).

STUDY DESIGN. The investigators have designed a prospective, multicentre, open-label clinical study that includes two multicentre randomized controlled trials (RCTs) based on the kidney biopsy report.

In the first RCT, patients with active renal lesions (E1 and/or C1), daily proteinuria >0.5 g and GFR ≥ 30 ml/min/1.72 m2 will be enrolled. They will be randomized to receive corticosteroids combined with RASBs in the experimental arm or RASBs alone in the control arm. Aim of this trial is to demostrate the benefit of corticosteroids in patients with active renal lesions.

In the second RCT, patients with chronic renal lesions (T1,2) and patients with moderate renal lesions (M0,1; S0,1; T0; E0; C0) at high or very high CKD risk (proteinuria> 0.5 g/day and GFR ≥ 30ml/min/1.73 m2) will be enrolled. They will be randomized to receive SGLT2 inhibitor (SGLT2i) combined with RASBs (experimental arm) or RASBs combined with corticosteroids (control arm). Aim of this trial is demostrate the benefit of SGLT2i combined with RASBs.

In conclusion, we have designed two RCTs (i) to study personalized therapy in biopsy-proven IgAN patients and (II) to monitor the outcomes to look at whether personalized therapy may delay the time to reach the ESKD predicted by our IgAN tool.

RECRUITMENT AND FOLLOW-UP. Renal Units will be involved in the enrollment of IgAN patients during a period of three years. The follow-up study to measure the outcomes will consist of regular visits at the prescribed times and to collect clinical and laboratory data and information on drug adherence. At the end of the trial, each patient will receive a final visit in the outpatient section.

OTHER MEAUSURES. Age, body mass index, eradication of infectious foci, or concurrent antibiotic therapy to prevent infections or to avoid the transformation of a trivial infection into a severe complication will be considered. Covid-19 vaccination will be done in all patients who will receive corticosteroids therapy. In addition, home and life conditions and culture will be analyzed. Regular daily exercise to prevent obesity and cardiovascular disease will be prescribed.

Dietary counseling. Patients with CKD stage 1 and 2 will observe the Mediterranean diet combined with reduced intake of proteins (1.0 - 0.8 g/kg bw/day). A reduced intake of proteins (0.6 - 0.8 g/kg bw/day) will also be prescribed to patients with CKD stage 3. Salt intake will be limited to 1.5 g/day. Dietary compliance will be assessed by measuring daily urinary sodium and urea excretion. Physical activity will be observed for 30 min. every day, primarily in the morning.

Severe adverse events. Infections, impaired glucose tolerance, weight gain, hypoglycemia will be monitored during the follow-up.

VARIABLES OF THE DISEASE. Kidney biopsy will be scored according to the Oxford classification because it is a simple method for predicting renal outcomes and for differentiating active and chronic renal lesions. Therefore, the kidney biopsy will be the principal key-note, not only for diagnosis but also for personalized therapy, because active renal lesions will be treated with immediate corticosteroid therapy before lesions become chronic. In some RCTs IgAN patients received six months of RASBs treatment before their enrollment for corticosteroid therapy. In our opinion this approach is not correct because the acute renal lesions evolve in the chronic stage and are no-responsive to corticosteroid therapy. Therefore, the aim of the first RCT is early treatment of the active renal lesions because they are responsible for altered GFR and proteinuria.

The definition of remission or no response of the MESTC lesions to therapy in published studies is inconsistent. Therefore, high-quality clinical trials with a large sample size are necessary to define the response of histological renal lesions to corticosteroids in biopsy-proven IgAN. The kidney biopsy will be analyzed using digital histopathologic analysis coupled with machine-learning tools. At least eight glomeruli will be available for a correct diagnosis. Renal tissue sections will be stained with hematoxylin and eosin, periodic acid-Schiff and methenamine silver. The last edition of the Oxford classification (MESTC) will be used for scoring the renal lesions.

Three independent renal pathologists, blinded to the study results, will score the lesions in the kidney biopsy using the Aperio System. The histology report will be necessary for the enrollment of patients. No larger RCT has confirmed that the disease improves when clinical decisions are made in a short time in the presence of the MESTC score.

* Serum creatinine will be measured using enzymatic methods calibrated to the National Institute of Standards and Technology's (NIST) liquid chromatography isotope dilution mass spectrometry method. eGFR creatinine will be evaluated by the CKD-EPI formula. Moreover, the slope of eGFR (16) will be calculated. Patients, categorized in CKD stages 1 to 3, will be included in the clinical study.
* Proteinuria. Patients will collect 24 hour urine for proteinuria. Values of >0.5 g/ day will be considered abnormal. Proteinuria reduction (geometric mean of 30% within 6 months), time-average proteinuria (TA-P) and slope of proteinuria will be evaluated.

Serum creatinine, proteinuria, age and hypertension have a lower weight when histological lesions are not considered. This finding highlights the importance of the kidney biopsy, not only for diagnosis but for personalized treatment.

* Blood hypertension is defined when values are > 130/80 mmHg or in subjects treated with anti-hypertensive drugs.
* For hyperuricemia allopurinol therapy is recommended.

SAMPLE SIZE CALCULATION.

ACIgAN. Data from the literature show a difference in renal survival between corticosteroids and controls when the researchers assumed a difference of 50% in the primary end point (i.e. in the between-arms difference of delta 24 hour proteinuria from baseline to 6 months) as clinically relevant. We assume that a mean delta proteinuria (±SD) from baseline to 6 months in patients treated with Ramipril alone (control arm) is 0.6±1.0 g/24 hours versus a mean delta proteinuria (±SD) from baseline to 6 months in patients treated with Ramipril and corticosteroids (experimental arm) 1.2±1.0 g/24 hours. Based on these assumptions, we calculated a sample size of 132 patients (66 patients per group including a 10% dropout rate) for a power of 90%, a two-sided significance level of 0.05 and 3 years of recruitment. If the number of the enrolled patients will be insufficient, the recruitment period will be extended for two years. At 4 months, all patients of the control arm who will display a 24 hour proteinuria >0.5g will be switched to the experimental treatment and will receive corticosteroids combined with RASBs for 4 months. They will be followed-up until the study termination.

CHRONIgAN. Data from the literature suggest a difference of renal survival between SGLT2is and controls. Here we assume a difference of 40% in the primary end point (i.e. in the between-arms difference of delta 24 hour proteinuria from baseline to 6 months) as clinically relevant. We assume that a mean delta proteinuria (±SD) from baseline to 6 months in patients with Ramipril alone is 0.6±1.0 g/24 hours versus a mean delta proteinuria (±SD) from baseline to 6 months in patients treated with SGLT-2 inhibitor and Ramipril (1.0±1.0 g/24 hours). Based on these assumptions, we have calculated a sample size of 294 patients (147 patients per group including a 10% dropout rate) for a power of 90%, a two-sided significance level of 0.05 and 3 years of recruitment. If the time-recruitment will be insufficient, the recruitment period will be extended for two years. At 6 months, all patients of the control arm who will display a 24 hour proteinuria >0.5 g will be switched to the experimental treatment (SGLT-2 inhibitor combined with Ramipril). They will be followed-up until the study termination.

ELIGIBILITY:
Inclusion Criteria:

* Only adult patients (age 18-70 years) with biopsy-proven idiopathic IgAN.
* IgAN patients with active or chronic or moderate renal lesions

Exclusion Criteria

* Patients with idiopathic IgAN and nephrotic syndrome (minimal change disease at kidney biopsy)
* IgAN patients with hematuria and acute renal failure
* IgAN patients with rapidly progressive glomerulonephritis (extracapillary lesions in more than 50% of glomeruli)
* Patients with secondary IgAN (lupus nephritis, Schoenlein-Henoch purpura, liver cirrhosis)
* Any prior immunosuppressive therapy
* Superimposed IgAN in kidney transplant
* Severe liver diseases
* Infections
* Malignancies
* Pregnancy
* Patients with myocardial infarction or cerebrovascular stroke in the previous 6 months
* Uncontrolled diabetes
* Aseptic necrosis of any bone
* Other conditions that can be exacerbated by corticosteroids
* Previous adverse side effects to RASBs
* Previous adverse side effects to SGLT2is
* Patients with mild renal lesions (M0,E0,S0,T0,C0), minor urinary findings, proteinuria < 0.5 g/day, normal GFR and normal blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
-Proteinuria reduction within 6 months in IgAN patients with active renal lesions | 6th month
  Reduction of proteinuria will be calculated as difference betweeen arms within 6 months
Proteinuria reduction within 6 months in IgAN patients with active renal lesions | 12th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN patients with active renal lesions | 18th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN patients with active renal lesions | 24th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN patients with active renal lesions | 30th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN patients with active renal lesions | 36th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN patients with chronic renal lesions | 6th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN patients with chronic renal lesions | 12th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN with chronic renal lesions | 18th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN patients with chronic renal lesions | 24th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN with chronic renal lesions | 30th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months
Proteinuria reduction within 6 months in IgAN with chronic renal lesions | 36th month
  Reduction of proteinuria will be calculated as difference betweeen arms within every 6 months

SECONDARY OUTCOMES:
eGFR slope change in IgAN patients with active renal lesions | 6th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with active renal lesions | 12th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with active renal lesions | 18th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with active renal lesions | 24th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with active renal lesions | 30th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with active renal lesions | 36th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with chronic renal lesions | 6th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with chronic renal lesions | 12th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with chronic renal lesions | 18th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with chronic renal lesions | 24th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with chronic renal lesions | 30th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR slope change in IgAN patients with chronic renal lesions | 36th month
  eGFR slope change calculated as the mean of the individual slopes obtained from individual linear regression of eGFR over time;
eGFR decline >40% in IgAN patients with active renal lesions | 6th month
  eGFR decline >40% in IgAN patients with active renal lesions
eGFR decline >40% in IgAN patients with active renal lesions | 12th month
  eGFR decline >40% in IgAN patients with active renal lesions
eGFR decline >40% in IgAN patients with active renal lesions | 18th month
  eGFR decline >40% in IgAN patients with active renal lesions
eGFR decline >40% in IgAN patients with active renal lesions | 24th month
  eGFR decline >40% in IgAN patients with active renal lesions
eGFR decline >40% in IgAN patients with active renal lesions | 30th month
  eGFR decline >40% in IgAN patients with active renal lesions
eGFR decline >40% in IgAN patients with active renal lesions | 36th month
  eGFR decline >40% in IgAN patients with active renal lesions
eGFR decline >40% in IgAN patients with chronic renal lesions | 6th month
  eGFR decline >40% in IgAN patients with chronic renal lesions
eGFR decline >40% in IgAN patients with chronic renal lesions | 12th month
  eGFR decline >40% in IgAN patients with chronic renal lesions
eGFR decline >40% in IgAN patients with chronic renal lesions | 18th month
  eGFR decline >40% in IgAN patients with chronic renal lesions
eGFR decline >40% in IgAN patients with chronic renal lesions | 24th month
  eGFR decline >40% in IgAN patients with chronic renal lesions
eGFR decline >40% in IgAN patients with chronic renal lesions | 30th month
  eGFR decline >40% in IgAN patients with chronic renal lesions
eGFR decline >40% in IgAN patients with chronic renal lesions | 36th month
  eGFR decline >40% in IgAN patients with chronic renal lesions
composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with active renal lesions | 6th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with active renal lesions
composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with active renal lesions | 12th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with active renal lesions
composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with active renal lesions | 18th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with active renal lesions
composite endpoint: eGFR decline > 40%, ESKD and death due to kidney disease in IgAN patients with active renal lesions | 24th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with active renal lesions
composite endpoint: eGFR decline > 40%, ESKD and death due to kidney disease in IgAN patients with active renal lesions | 30th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with active renal lesions
composite endpoint: eGFR decline > 40%, ESKD and death due to kidney disease in IgAN patients with active renal lesions | 36th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with active renal lesions
composite endpoint: eGFR decline > 40%, ESKD and death due to kidney disease in IgAN patients with chronic renal lesions | 6th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with chronic rena lesions
composite endpoint: eGFR decline > 40%, ESKD and death due to kidney disease in IgAN patients with chronic renal lesions | 12th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with chronic rena lesions
composite endpoint: eGFR decline > 40%, ESKD and death due to kidney disease. in IgAN patients with chronic renal lesions | 18th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with chronic renal lesions
composite endpoint: eGFR decline > 40%, ESKD and death due to kidney disease. in IgAN patients with chronic renal lesions | 24th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with chronic renal lesions
composite endpoint: eGFR decline > 40%, ESKD and death due to kidney disease. in IgAN patients with chronic renal lesions | 30th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with chronic renal lesions
composite endpoint: eGFR decline > 40%, ESKD and death due to kidney disease. in IgAN patients with chronic renal lesions | 36th month
  composite endpoint: eGFR decline > 40%, ESKD (defined as long-term eGFR < 15 ml/min/1.73m2 for more than 3 months or need of maintenance dialysis or kidney transplantation) and death due to kidney disease in IgAN patients with chronic renal lesions
proteinuria reduction (geometric mean of 30% within 6 months) | 6th month
  proteinuria reduction in IgAN patients with chronic renal lesions
proteinuria reduction (geometric mean of 30% within 6 months) | 12th month
  proteinuria reduction in IgAN patients with chronic renal lesions
proteinuria reduction (geometric mean of 30% within 6 months) | 18th month
  proteinuria reduction in IgAN patients with chronic renal lesions
proteinuria reduction (geometric mean of 30% within 6 months) | 24th month
  proteinuria reduction in IgAN patients with chronic renal lesions
proteinuria reduction (geometric mean of 30% within 6 months) | 30th month
  proteinuria reduction in IgAN patients with chronic renal lesions
proteinuria reduction (geometric mean of 30% within 6 months) | 36th month
  proteinuria reduction in IgAN patients with chronic renal lesions
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with active renal lesions | 3rd month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with active renal lesions | 6th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with active renal lesions | 9th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with active renal lesions | 12th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with active renal lesions | 18th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with active renal lesions | 24th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with active renal lesions | 30th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with active renal lesions | 36th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with chronic renal lesions | 6th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with chronic renal lesions | 12th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with chronic renal lesions | 18th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with chronic renal lesions | 24th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with chronic renal lesions | 30th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement
time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement in IgAN patients with chronic renal lesions | 36 th month
  time-averaged proteinuria (TA-P) calculated as the weighted mean of all post-randomization measurement, with weights representing the time elapsed since the previous measurement

CONTACTS AND LOCATIONS:
Overall Officials: Francesco P Schena, Study Chair — Fondazione Schena; francesco P Schena, Study Director — Fondazione Schena
Locations (1):
- francesco paolo Schena, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other partners
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Six years
Access Criteria: Publications or reports
URL: http://www.fondazioneschena.org

REFERENCES:
- [Background] Schena FP, Nistor I. Epidemiology of IgA Nephropathy: A Global Perspective. Semin Nephrol. 2018 Sep;38(5):435-442. doi: 10.1016/j.semnephrol.2018.05.013. PMID 30177015
- [Background] Koyama A, Igarashi M, Kobayashi M. Natural history and risk factors for immunoglobulin A nephropathy in Japan. Research Group on Progressive Renal Diseases. Am J Kidney Dis. 1997 Apr;29(4):526-32. doi: 10.1016/s0272-6386(97)90333-4. PMID 9100040
- [Background] Manno C, Strippoli GF, D'Altri C, Torres D, Rossini M, Schena FP. A novel simpler histological classification for renal survival in IgA nephropathy: a retrospective study. Am J Kidney Dis. 2007 Jun;49(6):763-75. doi: 10.1053/j.ajkd.2007.03.013. PMID 17533019
- [Background] Chapter 10: Immunoglobulin A nephropathy. Kidney Int Suppl (2011). 2012 Jun;2(2):209-217. doi: 10.1038/kisup.2012.23. No abstract available. PMID 25018935
- [Background] Schena FP, Anelli VW, Trotta J, Di Noia T, Manno C, Tripepi G, D'Arrigo G, Chesnaye NC, Russo ML, Stangou M, Papagianni A, Zoccali C, Tesar V, Coppo R; members of the VALIGA study. Development and testing of an artificial intelligence tool for predicting end-stage kidney disease in patients with immunoglobulin A nephropathy. Kidney Int. 2021 May;99(5):1179-1188. doi: 10.1016/j.kint.2020.07.046. Epub 2020 Sep 2. PMID 32889014
- [Background] Working Group of the International IgA Nephropathy Network and the Renal Pathology Society; Roberts IS, Cook HT, Troyanov S, Alpers CE, Amore A, Barratt J, Berthoux F, Bonsib S, Bruijn JA, Cattran DC, Coppo R, D'Agati V, D'Amico G, Emancipator S, Emma F, Feehally J, Ferrario F, Fervenza FC, Florquin S, Fogo A, Geddes CC, Groene HJ, Haas M, Herzenberg AM, Hill PA, Hogg RJ, Hsu SI, Jennette JC, Joh K, Julian BA, Kawamura T, Lai FM, Li LS, Li PK, Liu ZH, Mackinnon B, Mezzano S, Schena FP, Tomino Y, Walker PD, Wang H, Weening JJ, Yoshikawa N, Zhang H. The Oxford classification of IgA nephropathy: pathology definitions, correlations, and reproducibility. Kidney Int. 2009 Sep;76(5):546-56. doi: 10.1038/ki.2009.168. Epub 2009 Jul 1. PMID 19571790
- [Background] Working Group of the International IgA Nephropathy Network and the Renal Pathology Society; Cattran DC, Coppo R, Cook HT, Feehally J, Roberts IS, Troyanov S, Alpers CE, Amore A, Barratt J, Berthoux F, Bonsib S, Bruijn JA, D'Agati V, D'Amico G, Emancipator S, Emma F, Ferrario F, Fervenza FC, Florquin S, Fogo A, Geddes CC, Groene HJ, Haas M, Herzenberg AM, Hill PA, Hogg RJ, Hsu SI, Jennette JC, Joh K, Julian BA, Kawamura T, Lai FM, Leung CB, Li LS, Li PK, Liu ZH, Mackinnon B, Mezzano S, Schena FP, Tomino Y, Walker PD, Wang H, Weening JJ, Yoshikawa N, Zhang H. The Oxford classification of IgA nephropathy: rationale, clinicopathological correlations, and classification. Kidney Int. 2009 Sep;76(5):534-45. doi: 10.1038/ki.2009.243. Epub 2009 Jul 1. PMID 19571791
- [Background] Kang SH, Choi SR, Park HS, Lee JY, Sun IO, Hwang HS, Chung BH, Park CW, Yang CW, Kim YS, Choi YJ, Choi BS. The Oxford classification as a predictor of prognosis in patients with IgA nephropathy. Nephrol Dial Transplant. 2012 Jan;27(1):252-8. doi: 10.1093/ndt/gfr295. Epub 2011 May 23. PMID 21606384
- [Background] Rauen T, Eitner F, Fitzner C, Sommerer C, Zeier M, Otte B, Panzer U, Peters H, Benck U, Mertens PR, Kuhlmann U, Witzke O, Gross O, Vielhauer V, Mann JF, Hilgers RD, Floege J; STOP-IgAN Investigators. Intensive Supportive Care plus Immunosuppression in IgA Nephropathy. N Engl J Med. 2015 Dec 3;373(23):2225-36. doi: 10.1056/NEJMoa1415463. PMID 26630142
- [Background] Lv J, Zhang H, Wong MG, Jardine MJ, Hladunewich M, Jha V, Monaghan H, Zhao M, Barbour S, Reich H, Cattran D, Glassock R, Levin A, Wheeler D, Woodward M, Billot L, Chan TM, Liu ZH, Johnson DW, Cass A, Feehally J, Floege J, Remuzzi G, Wu Y, Agarwal R, Wang HY, Perkovic V; TESTING Study Group. Effect of Oral Methylprednisolone on Clinical Outcomes in Patients With IgA Nephropathy: The TESTING Randomized Clinical Trial. JAMA. 2017 Aug 1;318(5):432-442. doi: 10.1001/jama.2017.9362. PMID 28763548
- [Background] Shen XH, Liang SS, Chen HM, Le WB, Jiang S, Zeng CH, Zhou ML, Zhang HT, Liu ZH. Reversal of active glomerular lesions after immunosuppressive therapy in patients with IgA nephropathy: a repeat-biopsy based observation. J Nephrol. 2015 Aug;28(4):441-9. doi: 10.1007/s40620-014-0165-x. Epub 2015 Jan 14. PMID 25585823
- [Background] Shi SF, Wang SX, Jiang L, Lv JC, Liu LJ, Chen YQ, Zhu SN, Liu G, Zou WZ, Zhang H, Wang HY. Pathologic predictors of renal outcome and therapeutic efficacy in IgA nephropathy: validation of the oxford classification. Clin J Am Soc Nephrol. 2011 Sep;6(9):2175-84. doi: 10.2215/CJN.11521210. Epub 2011 Aug 18. PMID 21852672
- [Background] Lv J, Yang Y, Zhang H, Chen W, Pan X, Guo Z, Wang C, Li S, Zhang J, Zhang J, Liu L, Shi S, Wang S, Chen M, Cui Z, Chen N, Yu X, Zhao M, Wang H. Prediction of outcomes in crescentic IgA nephropathy in a multicenter cohort study. J Am Soc Nephrol. 2013 Dec;24(12):2118-25. doi: 10.1681/ASN.2012101017. Epub 2013 Sep 12. PMID 24029421
- [Background] Trimarchi H, Barratt J, Cattran DC, Cook HT, Coppo R, Haas M, Liu ZH, Roberts IS, Yuzawa Y, Zhang H, Feehally J; IgAN Classification Working Group of the International IgA Nephropathy Network and the Renal Pathology Society; Conference Participants. Oxford Classification of IgA nephropathy 2016: an update from the IgA Nephropathy Classification Working Group. Kidney Int. 2017 May;91(5):1014-1021. doi: 10.1016/j.kint.2017.02.003. Epub 2017 Mar 22. PMID 28341274
- [Background] Levey AS, Eckardt KU, Dorman NM, Christiansen SL, Hoorn EJ, Ingelfinger JR, Inker LA, Levin A, Mehrotra R, Palevsky PM, Perazella MA, Tong A, Allison SJ, Bockenhauer D, Briggs JP, Bromberg JS, Davenport A, Feldman HI, Fouque D, Gansevoort RT, Gill JS, Greene EL, Hemmelgarn BR, Kretzler M, Lambie M, Lane PH, Laycock J, Leventhal SE, Mittelman M, Morrissey P, Ostermann M, Rees L, Ronco P, Schaefer F, St Clair Russell J, Vinck C, Walsh SB, Weiner DE, Cheung M, Jadoul M, Winkelmayer WC. Nomenclature for kidney function and disease: report of a Kidney Disease: Improving Global Outcomes (KDIGO) Consensus Conference. Kidney Int. 2020 Jun;97(6):1117-1129. doi: 10.1016/j.kint.2020.02.010. Epub 2020 Mar 9. PMID 32409237
- [Background] Orlandi PF, Xie D, Yang W, Cohen JB, Deo R, Ricardo AC, Schrauben S, Wang X, Hamm LL, He J, Sondheimer JH, Kallem K, Townsend R, Raj D, Parsa A, Anderson AH, Feldman HI; CRIC Study Investigators; Chronic Renal Insufficiency Cohort (CRIC) Study Investigators. Slope of Kidney Function and Its Association with Longitudinal Mortality and Cardiovascular Disease among Individuals with CKD. J Am Soc Nephrol. 2020 Dec;31(12):2912-2923. doi: 10.1681/ASN.2020040476. Epub 2020 Oct 6. PMID 33023926
- [Background] Reich HN, Troyanov S, Scholey JW, Cattran DC; Toronto Glomerulonephritis Registry. Remission of proteinuria improves prognosis in IgA nephropathy. J Am Soc Nephrol. 2007 Dec;18(12):3177-83. doi: 10.1681/ASN.2007050526. Epub 2007 Oct 31. PMID 17978307
- [Background] Lea J, Greene T, Hebert L, Lipkowitz M, Massry S, Middleton J, Rostand SG, Miller E, Smith W, Bakris GL. The relationship between magnitude of proteinuria reduction and risk of end-stage renal disease: results of the African American study of kidney disease and hypertension. Arch Intern Med. 2005 Apr 25;165(8):947-53. doi: 10.1001/archinte.165.8.947. PMID 15851648
- [Background] Levin A, Agarwal R, Herrington WG, Heerspink HL, Mann JFE, Shahinfar S, Tuttle KR, Donner JA, Jha V, Nangaku M, de Zeeuw D, Jardine MJ, Mahaffey KW, Thompson AM, Beaucage M, Chong K, Roberts GV, Sunwold D, Vorster H, Warren M, Damster S, Malik C, Perkovic V; participant authors of the International Society of Nephrology's 1st International Consensus Meeting on Defining Kidney Failure in Clinical Trials. International consensus definitions of clinical trial outcomes for kidney failure: 2020. Kidney Int. 2020 Oct;98(4):849-859. doi: 10.1016/j.kint.2020.07.013. PMID 32998816
- [Background] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] El Karoui K, Fervenza FC, De Vriese AS. Treatment of IgA Nephropathy: A Rapidly Evolving Field. J Am Soc Nephrol. 2024 Jan 1;35(1):103-116. doi: 10.1681/ASN.0000000000000242. Epub 2023 Sep 29. PMID 37772889